CLINICAL TRIAL: NCT03252093
Title: A Randomized, Placebo-controlled, Double Blind Evaluation of the Safety and Efficacy of Angiotensin 1-7 (Ang-(1-7)) to Enhance Cognitive Function in Participants Undergoing Coronary Artery Bypass Graft (CABG) Surgery.
Brief Title: Evaluation of the Safety and Efficacy of Ang-(1-7) to Enhance Cognitive Function in Participants Undergoing CABG
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Funding ended
Sponsor: University of Arizona (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Suburban Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HL131014; 1U01HL131014-01A1 (NIH)
Record Dates: First submitted 2017-08-01; First posted 2017-08-17 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Coronary Artery Bypass Surgery; Cognitive Impairment
MeSH Terms: conditions — Cognitive Dysfunction | interventions — angiotensin I (1-7)

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Angiotensin-(1-7) (Experimental): Intervention: Drug: 200 mcg/kg/day injected subcutaneously once daily for 21 days
  Interventions: Drug: Angiotensin-(1-7)
- Placebo for Angiotensin-(1-7) (Placebo Comparator): Intervention: Placebo for Angiotensin-(1-7) injected subcutaneously once daily for 21 days
  Interventions: Drug: Placebo for Angiotensin-(1-7)

INTERVENTIONS:
Drug: Angiotensin-(1-7) — Subcutaneous injection of 200 mcg/kg/day
  Arms: Angiotensin-(1-7)
Drug: Placebo for Angiotensin-(1-7) — Subcutaneous injection of Placebo
  Arms: Placebo for Angiotensin-(1-7)

SUMMARY:
Coronary Artery Bypass Graft (CABG) is a surgical procedure known to be associated with cognitive impairment. Mechanisms of cognitive impairment are complex but may include insufficient oxygenation and inflammation due to exposure to the bypass circuit. Currently there are no approved therapeutics for the prevention or treatment of cognitive impairment in these patients.

A small peptide, Angiotensin-(1-7) [Ang-(1-7)], is known to decrease inflammation in the brain in animal models. Early studies in humans have shown it to be safe. This peptide is naturally produced by the body and has anti-inflammatory and vasodilatory effects. Investigators believe that Ang-(1-7) may be able to help lower the risk of cognitive dysfunction in patients undergoing CABG.

The goal of this project is to explore effects of the experimental peptide Angiotensin-(1-7) (Ang-(1-7) in patients undergoing an elective CABG surgery to determine its safety and efficacy to prevent cognitive dysfunction in patients undergoing CABG.

DETAILED DESCRIPTION:
Up to 104 participants (ages 60-80) undergoing elective CABG surgery at the Banner University Medical Center in Tucson, AZ or at Suburban Hospital/NIH Clinical Center in Bethesda, MD, will be enrolled in this randomized, placebo-controlled, double-blind study of Angiotensin-(1-7). Subjects who have a pre-operative neurologic, learning or psychiatric disorder will be excluded. In addition, a concurrent group of 20 age-matched adults will be recruited as a neuropsychological control group and will undergo neuropsychological testing at baseline, Day 21 and Day 90.

Participants will be asked to undergo a screening process to confirm eligibility and to rule out depression, dementia and contraindications to MRI. Prior to randomization, baseline measures will include neuropsychological testing, brain MRI, quality of life questionnaires, inflammatory markers and DNA/RNA sample collection. Participants will be treated for 21 days with a daily dose of subcutaneous Ang-(1-7) (100 mcg/kg/day) (n=60) or placebo (n=30). These measures will then be repeated at Day 21 and Day 90. The MRI will be repeated at Day 21 only.

Pharmacokinetic measurements will be obtained prior to administration of Ang-(1-7) or placebo and hourly for 6 hours following the first 6 doses. Delirium testing will occur on a daily basis post surgery until discharge. Serum study drug level will be obtained at Day 21.

Lastly, subjects will be followed on a weekly basis by telephone for all 12 weeks of the study.

1. Primary Objective: To evaluate the safety and tolerability of 21 days of subcutaneous (s.c.) once daily administration of Ang-(1-7) in eligible participants undergoing first-time, elective coronary artery bypass graft (CABG) surgery.
2. Secondary Objectives:

   1. To determine the pharmacokinetics of 21 days of treatment with Ang-(1-7).
   2. To determine if 21 days of treatment with 200 mcg/kg/day of Ang-(1-7) improves memory function measured as a change in performance from baseline to follow up on a composite score comprised of memory, executive functioning, language and processing speed in Ang-(1-7) treatment group compared to placebo controls and non-surgical controls.
   3. To determine if treatment with 200 mcg/kg/day Ang-(1-7) decreases postoperative delirium length and severity as measured with the Confusion Assessment Method (CAM) D2 to D7 ( or discharge) after surgery as compared to treatment with placebo group.
   4. To determine if 21 days of treatment with 200 mcg/kg/day Ang-(1-7) improves participant self-reported outcomes using standardized Kansas City Cardiomyopathy Questionnaire (KCCQ) and Instrumental Activities of Daily Living (IADL) measurement tools.
   5. To determine if 21 days treatment with 200 mcg/kg/day Ang-(1-7) results in changes in suicidal ideation and behavior as assessed by The Columbia Suicide Severity Rating Scale (C-SSRS).
   6. To compare postoperative mortality and morbidity at 90 days in the 200 mcg/kg/day Ang-(1-7) treatment group with the placebo group.
   7. To determine if 21 days of treatment of 200 mcg/kg/day Ang-(1-7) decreases postoperative observable changes in brain fractional anisotropy as measured by diffuse on magnetic resonance imaging (MRI) as compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

* Adult male or female first time cardiac surgical participants
* Elective on pump coronary artery bypass grafting (CABG)
* Age 60-80
* Signed, informed consent
* Geriatric Depression Scale score less than or = 14or Beck's Depression Inventory less than or = 20
* Score > or = 25 on the Mini-Mental State Examination (MMSE)

Exclusion Criteria:

* Recent (within 60 days) Cerebrovascular disease with neurological change
* Malignancy or pre-malignant state within 5 years not including non-melanoma skin cancer
* History of liver dysfunction with ongoing sequelae (including but not limited to liver enzymes > 2.5 x upper limit or normal (ULN) at screening).
* History of renal dysfunction with ongoing sequelae (including but not limited to creatinine value > 2.5 mg/dL at screening).
* Significant Lung Disease (FEV1< 1.5 L, pO2 <70 on room air, pCO2 >45)
* Presence of any severe mental illness that could affect interpretation of efficacy data, such as schizophrenia or bipolar affective disorder; any untreated or unstable psychiatric condition including depressive disorder or anxiety disorder.
* Active substance abuse
* Less than Grade 7 education or inability to read and perform cognitive assessment.
* Significant neurological disorder affecting memory
* Uncontrolled atrial fibrillation prior to surgery
* Concurrent use of prescription medications specifically for memory enhancement including herbal or natural supplements
* General anesthesia (defined as anesthesia requiring intubation or ventilatory support) within 3 months prior to randomization.
* Cardiopulmonary bypass or thoracotomy within 2 years prior to randomization.
* Chronic obstructive pulmonary disease (COPD) requiring oxygen therapy.
* Participants on immunosuppressive drugs, such as azathioprine, chemotherapeutic agents, mycophenolate, monoclonal antibodies, or more than 20 mg/day prednisone, within the previous 3 months
* Receipt of any investigational agent or device within 30 days of screening
* MRI contraindication not limited to abnormally high weight or height to fit in scanner (Bore 70cm); Presence of device/hardware incompatible with MR imaging
* Conditions causing severe anemia
* Participant is practicing Jehovah Witness
* Sexually active males not practicing a medically acceptable method of contraception, unless there is documented azoospermia.

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2017-07-20 (Actual); Primary Completion 2022-11-15 (Actual); Study Completion 2022-11-15 (Actual)

PRIMARY OUTCOMES:
Demonstrate 21 days daily administration of Ang-(1-7) in participants undergoing 1st time CABG surgery is safe and efficacious as assessed by the number of related AEs grade 3 or > and change in composite neuropsychological score up to Day 90. | Up to Day 90
  Adverse events (AEs), including serious adverse events (SAEs) will be monitored from the time of enrollment through Day 90. The number of AEs, withdrawals due to AE, and withdrawals for other reasons will be tabulated. Additional assessments include: serum blood levels of the Ang-(1-7) at Day 1, Day 3, Day 5 or Discharge and Day 21. Lastly blood pressuring monitoring pre and post treatment will occur Day 1 to discharge.
  Change in performance on composite scores of memory, executive functioning, language and processing speed in the treatment arm compared to placebo arm and non-surgical controls measured at 3 time points will assess the effectiveness of Ang-(1-7) in reducing postoperative cognitive impairment in CABG patients.

SECONDARY OUTCOMES:
Demonstrated change in the neuropsychological component scores assessed at baseline, Day 21 and Day 90 in the treatment and placebo arms. | Up to Day 90
  The component scores to be analyzed will include Rey Auditory Verbal Learning Test (RAVLT) and Confusion Assessment Method (CAM), assessment of general intellectual functioning (North American Adult Reading Test), prospective memory (MIST; Memory Intentions Test) , Visual Paired Associates, Object-Spatial Locations, three areas of executive functions including updating (Keep Track), shifting (Letter-Number), and inhibition (Stroop Color-Word), and psychomotor speed (Deary Simple and Complex Reaction Times, Trials A and B).
Evidence of change in fractional anisotropy from diffusion tensor imaging on Brain MRI at baseline versus post operative Day 21 will be assessed in the treatment and placebo arms as a measure of efficacy. | Up to Day 21
  CABG surgery will result in observable changes in gray matter volumes and integrity of white matter as measured by structural and diffusion MR imaging in all participants. Similar voxel-based multivariate regression analyses will be used for other MRI measures including gray and white matter volumes, axial and radial diffusion, and ASL perfusion. Comparisons between CABG patients and controls will use the general linear model in SPM8 with group (CABG, controls) as a categorical factor and age as a mean-centered control variable. For structural MRI, ICV will also be included as a covariate.
Demonstrated change in PBR28 VT/fP, a quantitative measure of TSPO receptor density, in a composite cerebral region-of-interest (ROI) derived from brain PET imaging in the treatment and placebo arms. | Up to Day 21
  PBR28 VT/fP will be measured in a composite cerebral region-of-interest (ROI), including automatic anatomically labeled, bilateral medial and lateral temporal, parietal, precuneus, prefrontal ROIs (Reiman, 2009) in the treatment and placebo arms.
Demonstrated associations between neuropsychogical test results, MRI findings and PBR28 binding in all participants. | Up to Day 90
  Neuropsychological testing outcomes and MRI findings will analyzed to evaluate associations between these outcomes and PBR28 binding. In addition, systemic inflammatory markers will be measured, including GM-CSF, IFNγ, IL-1 β, IL-2, IL-4, IL-5, IL-6, IL-7, IL-8, IL-10, IL-12 (p70), IL-13, and TNFα.

CONTACTS AND LOCATIONS:
Overall Officials: Nancy K Sweitzer, MD, PhD, Principal Investigator — University of Arizona
Locations (5):
- United States (5):
  - Banner- University Medical Center Phoenix, Phoenix, Arizona
  - University of Arizona Sarver Heart Center, Tucson, Arizona
  - Suburban Hospital, Bethesda, Maryland
  - National Institutes of Health, Bethesda, Maryland
  - INOVA Heart & Vascular Research, Falls Church, Virginia